CLINICAL TRIAL: NCT01776372
Title: Effect of the Use of a Digital Pleural Drainage System on Reducing Pleural Effusion Formation Following Lung Resection
Brief Title: Comparison of Pleural Drainage Systems on Reducing Pleural Effusion Formation Following Lung Resection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: SJHHPleuralDrainageComparsion; R.P. 12-3800 (Other: Hamilton Integrated Research Ethics Board)
Record Dates: First submitted 2013-01-21; First posted 2013-01-28 (Estimated); Last update posted 2014-05-13 (Estimated); Status verified 2014-05

CONDITIONS: Lung Neoplasms; Pleural Effusion
Keywords: Drainage; Chest tubes; Randomized Controlled Trial
MeSH Terms: conditions — Lung Neoplasms; Pleural Effusion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Digital thoracic drainage system (Active Comparator): Medela Thopaz Thoracic Drainage System
  Interventions: Device: Medela Thopaz Thoracic Drainage System
- Non-digital thoracic drainage system (Active Comparator): Atrium Express Dry Seal Chest Drain
  Interventions: Device: Atrium Express Dry Seal Chest Drain

INTERVENTIONS:
Device: Medela Thopaz Thoracic Drainage System
  Arms: Digital thoracic drainage system
Device: Atrium Express Dry Seal Chest Drain
  Arms: Non-digital thoracic drainage system

SUMMARY:
The chest cavity contains a small amount of fluid (pleural effusion). In normal circumstances this fluid is kept in balance. When surgery is performed on the lung, there can be accumulation of more fluid due to many causes. In order to drain this additional amount of pleural fluid, chest tube(s) are left in the thoracic cage after a lung resection procedure. The investigators are attempting to reduce the amount of pleural fluid production and formation by using a more balanced thoracic drainage system, which adjusts the amount of suction depending on the needs of the patient. That way, the amount of inflammation in the thoracic cage might be smaller, and hence less fluid will be formed. By this, the investigators are hoping that the chest tubes can be removed earlier, and the patients can be discharged faster and will potentially have a lower rate of re-admission to the hospital after surgery due to problems related to the fluid in the thoracic cage.

DETAILED DESCRIPTION:
Length of hospital stay after lung surgery depends mainly on duration of chest tube drainage. Patients undergoing lung resection have 1 or 2 chest tubes in the pleural cavity to evacuate air and pleural fluid. Digital drainage systems (recently approved for usage in Canada) offer the advantage of maintaining a stable intrapleural pressure through interactive balancing depending on the needs of the patient. In contrast, the traditional chest tube system offers continuous suctioning and negative pleural pressure, regardless the ongoing needs of the patients. Therefore, usage of digital drainage system (already shown to be beneficial in reducing the duration of air leak after lung resection when compared to the traditional system) may potentially reduce the amount of pleural drainage and hence reduce the duration of chest tube drainage until removal and overall patient's length of stay in hospital.

The following is a proposal for a randomized, controlled trial where patients will be randomized to have either a digital drainage system (intervention group) or non-digital drainage system, a conventional system currently used to drain the pleural space (the control group) after major lung resection for malignancy. The primary outcome of this study is comparing the overall amounts of pleural fluid drainage after major lung resection using two different chest tube drainage systems. Secondary outcomes will include measurement in time (hours) that chest tubes remain in-situ before removal following an operative procedure, and overall reduction in the length of stay (LOS) of patients; 90 days overall mortality and morbidity; occurrence of dyspnea related to the reoccurrence of pleural effusion; clinically significant reintervention needed (thoracocentesis, re-insertion of chest drain(s) and number and type of imaging studies required which are related to potential re-accumulation of pleural effusion); readmission rates within 1 month of discharge; comparison of pleural fluid/plasma protein ratio and inflammatory mediators (IL-6, IL-8, IL-10, IL-1RA, TNF-α) between the two groups, a potential indicator for differences in pleural inflammation and permeability between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be between 18 and 90 years of age
* Diagnosed with suspected lung cancer or metastatic cancer to the lungs
* Surgery must include lung resection (Wedge; single or multiple, lobectomy or bi-lobectomy) and mediastinal lymph nodes sampling or dissection
* Demonstrate an ability for understanding the study procedures
* Demonstrate willingness to remain on-study for the complete duration
* Must be able to give informed consent to participate at this study.

Exclusion Criteria:

* Patients undergoing lung resection due to non-malignancy
* Patients undergoing pneumonectomy
* Patients treated with neo-adjuvant chemotherapy and/or radiation prior to surgery
* Patients with previous lung resection on the ipsilateral side
* Patients with evidence of chronic heart failure (i.e. NYHA class III, IV; current treatment with diuretics for heart failure, and/or LVEF <35%)
* Patients with chronic renal failure (i.e. estimated CCr of < 50ml/min/m2)
* Patients with history of or ongoing liver disease, expressed by ascites or previous peritoneal tapping for ascites.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2013-01; Primary Completion 2013-08 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Overall quantity of pleural effusion (mL) | From one hour after surgery to chest tube removal, estimated duration of 3 days
  Overall amount of pleural effusion drained from patients undergoing lung resection until chest tubes removal, comparing the two systems. Fluid output will be measured and recorded every 8 hours, using a digital (Medela®) Thopaz drainage system or traditional non-digital Express (Atrium®) drainage system and the output will be recorded in milliliters. Chest tubes will be removed whenever the drainage is less than 350ml per 24 hours and when there is no active air leak

SECONDARY OUTCOMES:
Time chest tubes remain in-situ | An expected average of 3 days starting from transfer from OR
  Measurement of the time (in hours and days) that chest tubes remain in-situ following an operative procedure
Length of hospital stay | Estimated to be 4 days from admittance to discharge
Mortality and Morbidity | 90 days of surgery
  Overall mortality and morbidity
Occurrence of dyspnea related to the reoccurrence of pleural effusion | Estimated to be 4 days from admittance to discharge
Clinically significant reintervention needed | Estimated to be 4 days from admittance to discharge
  Clinically significant reintervention needed, including thoracocentesis, re-insertion of chest drain(s) and number and type of imaging studies required which are related to potential re-accumulation of pleural effusion
Readmission to hospital rates | Within 1 month of discharge
Comparison of pleural fluid/plasma protein ratio and inflammatory mediators | Samples to be taken in OR and on days 1, 2, 3 and 4 post-surgery
  Comparison of pleural fluid/plasma protein ratio and inflammatory mediators (IL-6, IL-8, IL-10, IL-1RA, TNF-α) between the two groups, a potential indicator for differences in pleural inflammation and permeability between the two groups

CONTACTS AND LOCATIONS:
Overall Officials: Yaron Shargall, MD FRCSC, Principal Investigator — McMaster University
Locations (1):
- St. Joseph's Healthcare Hamilton, Hamilton, Ontario, Canada